CLINICAL TRIAL: NCT00660946
Title: Correlation of Point of Care INR to Laboratory INR in Hemodialysis Patients Taking Warfarin
Brief Title: Comparison of Point of Care to Lab INR in Dialysis Patients on Warfarin
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Robert W. Hoel, Pharm D, Primary Investigator, Pharmacy Services Department, Mayo Clinic
Other Study IDs: 618-05
Record Dates: First submitted 2008-04-11; First posted 2008-04-17 (Estimated); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Anticoagulation in Dialysis Patients
Keywords: anticoagulation in dialysis patients; chronic anticoagulation; warfarin; hemodialysis; INR; Point of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 37 dialysis patients: 37 chronic hemodialysis patients on warfarin requiring Laboratory INR monitoring for anticoagulation management.

SUMMARY:
To determine whether point of care (POC) International Normalized Ratio (INR) test results correlate with plasma INR measures in hemodialysis patients.

DETAILED DESCRIPTION:
37 chronic hemodialysis patients being anticoagulated with warfarin require INR monitoring routinely.

ELIGIBILITY:
Inclusion Criteria:

* Chronic dialysis patients on chronic warfarin anticoagulation.

Exclusion Criteria:

* On warfarin for less than 1 month.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dialysis patients who undergo INR testing in the management their chronic warfarin therapy.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2005-06; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
To determine whether Point of Care INR testing would be suitable in the management of dialysis patients on chronic warfarin therapy | Not an intervention study, but observational in this cohort

SECONDARY OUTCOMES:
Determine whether Point of Care INR devices maintain test accuracy in dialysis patients who are temporarily anemic (HCT <32%) according to their CBC | Not an intervention study, but observational in the cohort (statistics completed 1.5 yrs)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W. Hoel, Pharm D, Principal Investigator — Mayo Clinic Rochester, Mn USA

REFERENCES:
- [Derived] Hoel RW, Albright RC, Beyer LK, Santrach PJ, Magtibay DL, Everson SL, McBane RD. Correlation of point-of-care International Normalized Ratio to laboratory International Normalized Ratio in hemodialysis patients taking warfarin. Clin J Am Soc Nephrol. 2009 Jan;4(1):99-104. doi: 10.2215/CJN.03360708. Epub 2008 Nov 5. PMID 18987294